CLINICAL TRIAL: NCT05945056
Title: Effectiveness of Frog Leg Technique in Management of Low Back Pain Due to Lumbar Lordosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Education Research Foundation (HERF) (Other)
Responsible Party: Principal Investigator, Mamoona Tasleem Afzal, Senior Lecturer, Health Education Research Foundation (HERF)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1309-PPDPT-008/ANAM JAVED
Record Dates: First submitted 2023-05-26; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain, Postural
Keywords: Low Back Pain; Frog Leg Technique; Exercise Therapy
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrotherapy with Frog Leg Exercise Intervention (Experimental): Experimental group received Frog leg technique along with transcutaneous electrical nerve stimulation for 10 sessions of duration half hour each on regular basis.
  Interventions: Other: Frog Leg Exercise; Other: Electrotherapy(Transcutaneous Electrical Nerve Stimulator)
- Standard Exercise Therapy with Electrotherapy (Active Comparator): Control group received standard exercise therapy treatment along with transcutaneous electrical nerve stimulation for 10 sessions of duration half hour each on regular basis.
  Interventions: Other: Electrotherapy(Transcutaneous Electrical Nerve Stimulator); Other: Exercise Therapy

INTERVENTIONS:
Other: Frog Leg Exercise — The patient lies supine with legs flexed, knees apart and the soles of the feet put together on couch. The physiotherapist stands at the side of the table, moves one arm between the legs to place the hand under the sacrum and cup it. The fingers spread to accommodate the spinous process of the fifth lumbar vertebra. The tips of the fingers contact and grasp the junction of the fifth lumbar vertebra and the base of the sacrum. This hand will give traction in a caudal direction throughout the procedure to move the sacral base posteriorly and the apex interiorly. patient is asked to take a deep breath and hold it, while at the same time they steadily slide the feet downward toward the end of the table.Then patient brings their legs back to the frog leg position, but as they do so the therapist maintains traction preventing the sacrum from moving cephalad. Procedure is repeated for a total of 8 repetitions.
  Arms: Electrotherapy with Frog Leg Exercise Intervention
Other: Electrotherapy(Transcutaneous Electrical Nerve Stimulator) — TENS or transcutaneous electrical nerve stimulator is a low voltage electric current to relieve pain. A small battery-operated TENS device which has leads connected to sticky pads called electrodes was used in treatment. Patient in lying position gets pads directly attached to skin of lumbar region. Small electrical impulses delivered to the affected area of the patient's body when the machine is switched on, which patient feel as a tingling sensation.
Other: Exercise Therapy — Stretching of tight muscles(hip flexors and lower back extensors) Abdominal Curl-Ups and Bridging exercises.
  Arms: Standard Exercise Therapy with Electrotherapy

SUMMARY:
Condition in which lumbar region experiences stress or extra weight and is arched to point of muscle pain or spasms is called Lumbar hyperlordosis.The study findings compared the effectiveness of frog leg technique and standard exercise therapy in management of low back pain due to lumbar lordosis.

DETAILED DESCRIPTION:
In adult population, a major health problem is Low back pain. Postural change is one of the risk factor. Abnormal posture causes strain on ligaments and muscles, as a result indirectly affects the curvature of the lumbar spine.Condition in which lumbar region experiences stress or extra weight and is arched to point of muscle pain or spasms is called Lumbar hyperlordosis.The study findings compared the effectiveness of frog leg technique and standard exercise therapy in management of low back pain due to lumbar lordosis.

ELIGIBILITY:
Inclusion Criteria:

* Females with age between 20 and 45 years
* Patients with low back ache due to lumbar lordosis

Exclusion Criteria:

* History of surgery
* Patients with discogenic backache.
* Backache in pregnancy.
* Patients with traumatic history.
* Patients with pain due to any reason other than lumbar lordosis.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females suffer more from lumbar lordosis,hence female participants were selected for study.
Enrollment: 28 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain | Data was Collected at Baseline, 5th Day & 10th Day.
  Visual Analogue Scale used to assess pain.
Change in Disability Level | Data was Collected at Baseline, 5th Day & 10th Day.
  Oswestry Low Back Pain Disability Questionnaire used to assess level of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Anam Javed, Master, Principal Investigator — Bashir Institute of Health Sciences

IPD SHARING:
Plan to Share IPD: No